CLINICAL TRIAL: NCT01081964
Title: A Phase 2, Multi-Dose, Double-Blind, Double-Dummy, Active-Control, Randomized Study to Evaluate the Safety, Efficacy and Pharmacokinetic Profile of Two Dosing Regimens of Zabofloxacin for the Treatment of Community-Acquired Pneumonia of Moderate Severity
Brief Title: Safety and Efficacy Study of Oral Zabofloxacin in Community Acquired Pneumonia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Financial considerations
Sponsor: IASO Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PB-101-200
Record Dates: First submitted 2010-02-19; First posted 2010-03-05 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Community Acquired Pneumonia
Keywords: pneumonia; Community acquired pneumonia of moderate severity
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — zabofloxacin; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Levofloxacin 500mg (Active Comparator): Levofloxacin 500mg once daily for 7 days
  Interventions: Drug: Levofloxacin 500mg
- Zabofloxacin 5 days (Experimental): Zabofloxacin 400mg for 5 days
  Interventions: Drug: Zabofloxacin 400mg
- Zabofloxacin 3 days (Experimental): Zabofloxacin 400mg for 3 days
  Interventions: Drug: Zabofloxacin

INTERVENTIONS:
Drug: Zabofloxacin — Zabofloxacin 400mg capsule once daily for 3 days
  Arms: Zabofloxacin 3 days
Drug: Levofloxacin 500mg — Levofloxacin 500mg orally for 7 days
  Arms: Levofloxacin 500mg
Drug: Zabofloxacin 400mg — Zabofloxacin 400mg orally for 5 days
  Arms: Zabofloxacin 5 days

SUMMARY:
A double-blind, three-arm study, to evaluate the safety and efficacy of two dosing regimens of zabofloxacin (a fluoroquinolone antibiotic) in community acquired pneumonia.

DETAILED DESCRIPTION:
The study is a Phase 2, global, prospective, multi-dose, double-blind, double-dummy, active-control, randomized, parallel-group, multicenter study of oral zabofloxacin HCl (400mg) versus oral levofloxacin (500mg) in the treatment of adults with community-acquired pneumonia of moderate severity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >/= 18 years old
* Documented fever (oral >100°F (37.8°C), tympanic >101°F (38.1°C)must be documented within the time frame of 24 hours prior to first dose through 24 hours after first dose of study drug
* Community-acquired pneumonia of moderate severity (defined as PSI Risk Class II or III) requiring administration of antibiotics
* Dyspnea and/or tachypnea (>20 breaths/minute)
* Clinical diagnosis of pneumonia, as demonstrated by all of the following signs and symptoms:

  1. new or increased cough
  2. production of purulent sputum or a change in the character of sputum in subjects who normally have purulent sputum
  3. auscultatory findings on pulmonary examination of rales and/or evidence of pulmonary consolidation (e.g., bronchial breath sounds, egophony, or dullness on percussion)
* Females must be surgically sterile (e.g., tubal ligation, hysterectomy), post-menopausal at least 2 years, or if of childbearing potential, they must have a negative urine pregnancy test (β-human chorionic gonadotropin [β-hCG]) prior to randomization into the study. Males and females must agree that if they have intercourse that they will use at least two medically accepted methods of birth control (e.g., hormonal contraceptive, intrauterine device, spermicide, or condom) from study entry through 60 days after discontinuation of study drug treatment
* Able to give written informed consent in a manner approved by the Institutional Review Board or Ethics Committee and comply with the requirements of the study

Exclusion Criteria:

Subjects must NOT meet any of the following exclusion criteria:

* Received one or more doses of any systemic antibiotic in the last 2 weeks
* Diagnosed with any other infection requiring systemic antibacterial therapy
* Require long-term (>7 days) antibiotic therapy
* Previous diagnosed condition that might mimic or complicate the course and evaluation of the infectious disease process (e.g., septic shock, bronchiectasis, lung abcess or empyema, aspiration pneumonia, active tuberculosis, pulmonary malignancy, cystic fibrosis, post-obstructive pneumonia, etc.)
* Hypothermia (oral <96°F [35.6°C}, tympanic <97°F [35.9°C]
* Hospitalization (inpatient) in the previous 60 days or infection presumably acquired in the hospital
* Resident of a skilled nursing facility anytime in the previous 60 days or infection presumably acquired in a skilled nursing facility
* Chronic infection with Hepatitis B
* Any evidence of, or is a known carrier of , Hepatitis C antibody
* Infection with Clostridium difficile
* Immunocompromising illness, including known human immunodeficiency virus (HIV) positivity or AIDS, organ (bone marrow) transplant recipients, and hematological malignancy
* Psychotic disease, peripheral neuropathy, and glucose-6-phosphate dehydrogenase deficiency; uncontrolled or poorly controlled diabetes. Diabetic subjects who are stable and on a stable course of antihyperglycemic agents for the past 3 months will be permitted in the trial.
* High exposure to sunlight or ultraviolet radiation
* Immunosuppressive therapy, including cancer chemotherapy or chronic use of corticosteroids (i.e., >20mg prednisone or equivalent per day for >/= 14 days within the last 6 months
* History of renal or hepatic disease as defined by at least one of the following:

  1. Calculated creatinine clearance <50 mL/min (any subject on dialysis must be excluded)
  2. BUN >/= 30 mg/dL
  3. ALT or AST > 3x ULN
  4. Total bilirubin > 2x ULN
  5. Alkaline phosphatase > 1.25x ULN
* History of or current malabsorption conditions (i.e., short bowel syndrome, active Crohn's disease, celiac disease, etc.)
* Neutropenia as defined by absolute neutrophil count <1000 cells/mm3. Subjects with neutrophil counts as low as 500 cells/mm3 are permitted if the reduction can be documented to be due to the acute infectious process
* Platelet count <75,000/mm3. Subjects with platelet counts as low as 50,000/mm3 are permitted if the reduction is historically stable
* Coagulation tests >1.5x ULN (PT, PTT, or INR). Subjects on anticoagulants with values > 1.5x ULN can be enrolled, provided these values are historically stable and within the therapeutic range
* History of alcohol or drug abuse in the past 2 years
* History of seizure or currently receiving anti-seizure medication anytime in the past year, or a seizure in the past year
* History of ventricular arrhythmia
* History of QTc prolongation (i.e., >450msec) or observed QTc measurement at screening > 450msec, or a history of additional risk factors for Torsade de Pointe, such as heart failure, hypokalemia, or familial history of Long QT syndrome
* Require medications that may prolong the QTc interval
* Require medications that affect absorption, including but not limited to sucralfate or cimetidine
* Require treatment with theophylline, probenecid, vitamin K antagonists (other than warfarin; subjects must be on stable dose of warfarin and within therapeutic range)
* Pregnant, planning to become pregnant, or breast feeding
* Received any investigational drug or device within 30 days prior to study entry
* Previously received zabofloxacin in a clinical trial
* History of allergy or intolerability to fluoroquinolones
* History of fluoroquinolone tendinopathy
* Evidence of immediately life-threatening disease including, but not limited to current or impending respiratory failure, acute heart failure, shock, acute coronary syndrome, unstable arrhythmias, hypertensive emergency, acute hepatic failure, active gastrointestinal bleeding, profound metabolic abnormalities (e.g., diabetic ketoacidosis), or acute cerebrovascular events
* Current condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the data
* Unable or unwilling to adhere to sthe study specified procedures and restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Safety | Up to 35 days after first dose
  Assess safety through monitoring of adverse events, ECGs, and the collection of conventional laboratory data (i.e., chemistry panel, CBC with differential, urinalysis)

SECONDARY OUTCOMES:
Efficacy of the two dosing regimens of zabofloxacin | Up to 35 days after first dose
  Determine the clinical response and microbiological response of two dosing regimens in the treatment of bacteriologically confirmed CAP of moderate severity; determine the pharmacokinetic profile in subjects with CAP.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Huntsville, Alabama
  - Toney, Alabama
  - Fort Myers, Florida
  - Eagle, Idaho
  - Evansville, Indiana
  - Keego Harbor, Michigan
  - Belvidere, New Jersey
  - Columbus, Ohio
  - Dayton, Ohio
  - Springfield, Ohio
  - Gresham, Oregon
  - Warminster, Pennsylvania
  - Tyler, Texas